CLINICAL TRIAL: NCT02762812
Title: International Multi-center Comparative Double-blind Randomized Clinical Trial to Evaluate Efficacy and Safety of BCD-055 (JSC "BIOCAD", Russia) and Remicade® in Patients With Ankylosing Spondylitis
Brief Title: Comparative Clinical Trial to Evaluate Efficacy and Safety of BCD-055 and Remicade® in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-055-2
Record Dates: First submitted 2016-04-04; First posted 2016-05-05 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — BCD-055; Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-055 (Experimental): Patients in this group will receive BCD-055 in a dose of 5 mg/kg on Week 0, Week 2, Week 6, Week 14, Week 22, Week 30, Wekk 38, Week 46, Week 54.
  Interventions: Biological: BCD-055
- Remicade® (Active Comparator): Patients in this group will receive Remicade® in a dose of 5 mg/kg on Week 0, Week 2, Week 6, Week 14, Week 22, Week 30, Wekk 38, Week 46, Week 54.
  Interventions: Biological: Remicade®

INTERVENTIONS:
Biological: BCD-055
  Other Names: infliximab
  Arms: BCD-055
Biological: Remicade®
  Other Names: infliximab
  Arms: Remicade®

SUMMARY:
BCD-055-2 is international multi-center comparative double-blind randomized clinical trial to evaluate efficacy and safety of BCD-055 (JSC "BIOCAD", Russia) and Remicade® in patients with ankylosing spondylitis.

BCD-055 is biosimilar of infliximab (JSC "BIOCAD", Russia)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Active ankylosing spondylitis according to modified criteria of New York classification (1984), that was diagnosed at least 3 months prior to screening.
* Active disease according to BASDAI (score 4 or more) if nonsteroidal antiinflammatory drugs were used in the last 3 month prior to screening.
* Mean backache intensity equals 4 points or more.

Exclusion Criteria:

* Previous therapy of ankylosing spondylitis with monoclonal antibodies (including tumor necrosis factor)
* Total spinal ankylosis
* History of tuberculosis
* Body mass more than 120 kg
* Patient is taking corticosteroids for up to 4 weeks in a dose more than 10 mg (recalculated to prednisolone) before signing informed consent.
* Prior use of disease-modifying antirheumatic drugs including methotrexate, sulfasalazin, chloroquine or hydroxychloroquine for up to 4 weeks before randomization.
* Prior use of alkylating agents for up to 12 months prior to signing informed consent.
* Intraarticular use of corticosteroids for up to 4 weeks before randomization.
* Prior use of live or attenuated vaccines for up to 8 weeks before signing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Ratio of patients with ASAS20 response after 30 weeks of therapy | Week 30
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more after 30 weeks of therapy with BCD-055.

SECONDARY OUTCOMES:
Ratio of patients with ASAS20 response after 14 and 54 weeks of therapy | Week 14, Week 54
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 20% or more after 14 and 54 weeks of therapy with BCD-055.
Ratio of patients with ASAS40 response after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Ratio of patients who developed a decrease in ankylosing spondylitis assessment score (ASAS) by 40% or more after 14, 30 and 54 weeks of therapy with BCD-055.
Mean change in BASDAI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) after 14, 30 and 54 weeks of therapy
Mean change in BASMI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean change in Bath Ankylosing Spondylitis Metrology Index (BASMI), after 14, 30 and 54 weeks of therapy
Mean change in BASFI after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean change in Bath Ankylosing Spondylitis Functional Index (BASFI) after 14, 30 and 54 weeks of therapy
Mean change in MASES after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) after 14, 30 and 54 weeks of therapy
Mean SF-36 score at screening and after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean score of quality of life as assessed by Short Form-36 (SF-36) at screening and after 14, 30 and 54 weeks of therapy
Mean chest excursion at screening and after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean chest excursion at screening and after 14, 30 and 54 weeks of therapy
Mean quantity of abnormal peripheral joints after 14, 30 and 54 weeks of therapy | Week 14, Week 30, Week 54
  Mean quantity of abnormal peripheral joints after 14, 30 and 54 weeks of therapy
Frequency of AE/SAE | 54 weeks
  Frequency of AE/SAE
Frequency of AE 3-4 grade CTCAE | 54 weeks
  Frequency of AE 3-4 grade CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (1):
- North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided